CLINICAL TRIAL: NCT00538824
Title: A Phase II Study of Dexamethasone (DECADRON®), Thalidomide (THALOMID®), and Lenalidomide (REVLIMID®) for Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Phase II Study of Dexamethasone, Thalidomide and Lenalidomide for Subjects With Relapsed or Refractory Multiple Myeloma
Acronym: DexTR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0708009381; RV-MM-PI-0132
Record Dates: First submitted 2007-10-02; First posted 2007-10-03 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Multiple Myeloma
Keywords: myeloma; relapsed or refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Recurrence | interventions — Dexamethasone; Thalidomide; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DexTR (all patients) (Experimental): All patients were treated with the DexTR (dexamethasone / thalidomide, lenalidomide (Revlimid®)), which consisted of lenalidomide 25mg/day during days 1-21, dexamethasone 40mg/day on days 1-4, 9-12, and 17-20, and thalidomide 50mg/day for the first 7 days, followed by 100mg/day for all subsequent days, for a total of 4 cycles of 28 days each.
  Interventions: Drug: dexamethasone; Drug: thalidomide; Drug: lenalidomide

INTERVENTIONS:
Drug: dexamethasone — Cycles 1-4 • Dexamethasone (40mg ) will be given on days 1-4, 9-12, 17-20 of a 28-day cycle.
  After completing 4 cycles:
  * Patients who demonstrate disease progression at any time will be taken off study.
  * Patients who achieve a resolution of monoclonal gammopathy as detected on serum immunofixation or achieve a plateau of disease (no change in M-spike as detected on serum protein electrophoresis) for > 2 cycles will be transitioned to maintenance therapy.
  * Patients who continue to respond without achieving either a plateau or a CR will continue on induction therapy until plateau for >2 cycles or CR in the absence of untoward toxicity. These patients will be then transitioned to maintenance therapy.
  Maintenance therapy will consist of:
  • Dexamethasone 20mg weekly days 1, 8, 15, 22 out of a 28 day cycle)
Drug: thalidomide — Cycles 1-4
  • Thalidomide will be given 50mg daily on days 1-7, thereafter 100mg daily on days 8-28 of the first 28-day cycle. Thalidomide will then be given at 100mg/daily for days 1-28 of each subsequent cycle.
  After completing 4 cycles:
  * Patients who demonstrate disease progression at any time will be taken off study.
  * Patients who achieve a resolution of monoclonal gammopathy as detected on serum immunofixation or achieve a plateau of disease (no change in M-spike as detected on serum protein electrophoresis) for > 2 cycles will be transitioned to maintenance therapy.
  * Patients who continue to respond without achieving either a plateau or a CR will continue on induction therapy until plateau for >2 cycles or CR in the absence of untoward toxicity. These patients will be then transitioned to maintenance therapy.
Drug: lenalidomide — Cycles 1-4 • Lenalidomide will be given 25mg daily for days 1-21 of each 28 day cycle.
  After completing 4 cycles:
  * Patients who demonstrate disease progression at any time will be taken off study.
  * Patients who achieve a resolution of monoclonal gammopathy as detected on serum immunofixation or achieve a plateau of disease (no change in M-spike as detected on serum protein electrophoresis) for > 2 cycles will be transitioned to maintenance therapy.
  * Patients who continue to respond without achieving either a plateau or a CR will continue on induction therapy until plateau for >2 cycles or CR in the absence of untoward toxicity. These patients will be then transitioned to maintenance therapy.
  Maintenance therapy will consist of:
  • Lenalidomide 25 mg/daily days 1 - 21 out of a 28 day cycle. 15mg/daily on days 1-21 of a 28 day cycle of lenalidomide will be given to patients with a creatinine clearance of < 40cc/min*

SUMMARY:
Study Objectives

1. To evaluate the efficacy of the combination of dexamethasone (Decadron®), thalidomide (Thalomid®), and lenalidomide (Revlimid®) as therapy for patients with relapsed or refractory multiple myeloma (MM) who have failed prior treatment with both lenalidomide and thalidomide when used as monotherapies.
2. To evaluate the safety of the combination of lenalidomide, dexamethasone, and thalidomide as a therapy for patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
This phase II study is a treatment program for patients with relapsed or refractory multiple myeloma who have had prior treatment with both thalidomide and lenalidomide in separate regimens each used as a single agent or in combination with corticosteroids. Up to 45 patients will be enrolled. Patients who sign informed consent form and RevAssist® and S.T.E.P.S® patient agreement form and fulfill all eligibility criteria will be enrolled.

DexTR therapy:

Cycles 1-4

* Dexamethasone (40mg ) will be given on days 1-4, 9-12, 17-20 of a 28-day cycle.
* Thalidomide will be given 50mg daily on days 1-7, thereafter 100mg daily on days 8-28 of the first 28-day cycle. Thalidomide will then be given at 100mg/daily for days 1-28 of each subsequent cycle.
* Lenalidomide will be given 25mg daily for days 1-21 of each 28 day cycle.
* Prophylactic medications, such as medications for thrombosis risk, will be given.

After completing 4 cycles:

* Patients who demonstrate disease progression at any time will be taken off study.
* Patients who achieve a resolution of monoclonal gammopathy as detected on serum immunofixation or achieve a plateau of disease (no change in M-spike as detected on serum protein electrophoresis) for > 2 cycles will be transitioned to maintenance therapy.
* Patients who continue to respond without achieving either a plateau or a CR will continue on induction therapy until plateau for >2 cycles or CR in the absence of untoward toxicity. These patients will be then transitioned to maintenance therapy.

Maintenance therapy:

Maintenance therapy will consist of:

* Dexamethasone 20mg weekly days 1, 8, 15, 22 out of a 28 day cycle)
* Lenalidomide 25 mg/daily days 1 - 21 out of a 28 day cycle. 15mg/daily on days 1-21 of a 28 day cycle of lenalidomide will be given to patients with a creatinine clearance of < 40cc/min*

  * Patients who finished induction therapy with DexTR at a reduced dose of lenalidomide will start maintenance therapy at the same dose of lenalidomide on which they ended induction therapy. For patients with a creatinine clearance of < 40cc / minute, the lenalidomide dose will be the lower of their last induction therapy dose or 15mg daily on days 1 - 21 out of a 28 day cycle.

Serial clinic visits and laboratory measurements will be performed to monitor for treatment response. Those patients who demonstrate progression of disease at any point during DexTR therapy will be taken off study.

At the end of every cycle (which may coincide with day 1 of the new cycle), response and toxicity will be evaluated. During cycle 1, patients will have lab work done weekly (CBC with differential and blood electrolytes). All patients will remain on study until disease progression or side effects become excessive. Patients who achieve a stable plateau and are on maintenance therapy as defined above may be taken off study if eligible to proceed to high dose chemotherapy and autologous stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Subject must voluntarily sign and understand written informed consent.
* Age > 18 years at the time of signing the consent form.
* Histologically confirmed Salmon-Durie stage II or III MM. Stage I MM patients will be eligible if they display poor prognostic factors (ß2M ≥5.5 mg/L, plasma cell proliferation index ≥5%, albumin of less then 3.0, and unfavorable cytogenetics).
* Relapsed or refractory myeloma as defined by Appendix II, table 1, progression of disease either after prior therapy or lack of response to currently used therapy.
* Prior treatment with prior lenalidomide and thalidomide as single agents or in combination with dexamethasone, but not in combination with each other.
* No anti-myeloma therapy within 14 days prior to initiation of study treatment. Patients may be receiving adjuvant antiresorptive therapy (i.e., pamidronate or zoledronic acid) as routine care.
* Measurable disease as defined by > 1.0 g/dL serum monoclonal protein, >0.1 g/dL serum free light chains, >0.2 g/24 hrs urinary M-protein excretion, and/or measurable plasmacytoma(s).
* Karnofsky performance status ≥70% (>60% if due to bony involvement of myeloma.
* All study participants must be registered into the mandatory RevAssist® and S.T.E.P.S.® programs, and be willing and able to comply with the requirements of the RevAssist® and S.T.E.P.S.® programs.
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of prescribing lenalidomide and thalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with females of child bearing potential even if they have had a successful vasectomy.
* Able to take aspirin daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).
* Life expectancy ≥ 3 months
* Subjects must meet the following laboratory parameters:

  * Absolute neutrophil count (ANC) ≥1000 cells/mm3 (1.0 x 109/L)
  * Platelets count ≥ 75,000/mm3 (75 x 109/L)
  * Serum SGOT/AST <3.0 x upper limits of normal (ULN)
  * Serum SGPT/ALT <3.0 x upper limits of normal (ULN)
  * Serum creatinine <2.5 mg/dL (221 µmol/L)
  * Serum total bilirubin <2.0 mg/dL (34 µmol/L)

Exclusion Criteria:

* Patients with non-secretory MM (no measurable monoclonal protein, free light chains, and/or M-spike in blood or urine).
* Prior history of other malignancies (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless disease free for ≥ 5 years.
* Myocardial infarction within 6 months prior to enrollment , or NYHA(New York Hospital Association) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Pregnant or lactating females are ineligible.
* Given the potential of the study drugs to trigger or worsen HIV viremia and the incidence of opportunistic infections inpatients infected with the HIV virus, HIV-1 or HIV-2 positive patients will be excluded. The interactions of HAART with study drugs have not been determined.
* Active hepatitis B or hepatitis C infection.
* Active viral or bacterial infections or any coexisting medical problem that would significantly increase the risks of this treatment program.
* Any coexisting medical problem or laboratory evaluation that, in the treating physician's or principal investigator's opinion, makes the patient unsuitable to participate in this clinical trial.
* Known hypersensitivity to dexamethasone, lenalidomide, or thalidomide.
* History of thromboembolic event within the past 6 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2010-09-22 (Actual); Study Completion 2010-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Niesvizky, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- DexTR (All Patients): All patients were treated with the DexTR (dexamethasone / thalidomide, lenalidomide (Revlimid®)), which consisted of lenalidomide 25mg/day during days 1-21, dexamethasone 40mg/day on days 1-4, 9-12, and 17-20, and thalidomide 50mg/day for the first 7 days, followed by 100mg/day for all subsequent days, for a total of 4 cycles of 28 days each.
  dexamethasone: Cycles 1-4
  • Dexamethasone (40mg ) will be given on days 1-4, 9-12, 17-20 of a 28-day cycle.
  After completing 4 cycles:
  * Patients who demonstrate disease progression at any time will be taken off study.
  * Patients who achieve a resolution of monoclonal gammopathy as detected on serum immunofixation or achieve a plateau of disease (no change in M-spike as detected on serum protein electrophoresis) for > 2 cycles will be transitioned to maintenance therapy.
  * Patients who continue to respond without achieving either a plateau or a CR will continue on induction therapy until plateau for >2 cycles or CR in the absence of unt
Period: Overall Study
Arm/Group | DexTR (All Patients)
Started | 5
Progression of Disease | 2
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | DexTR (All Patients)
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 65 [50 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
serum creatinine at baseline (in mg/dL) [Median (Full Range); unit: mg/dL] | 3.8 [3.1 to 4.2]
Beta-2 microglobulin at baseline (in mg/L) [Median (Full Range); unit: mg/dL] | 4.1 [1.5 to 5.6]
lactage dehydrogenase at baseline (U/L) [Median (Full Range); unit: U/L] | 177 [150 to 225]
Durie-Salmon Classification [Number; unit: participants] — Subjects were staged according to the Durie salmon Staging Classification System. Criteria for the staging system can be found here: https://www.themmrf.org/multiple-myeloma/prognosis/myeloma-stages/durie-salmon-staging-system/.
  Staging classification describes multiple myeloma tumor burden; stage 1 is a low tumor burden/myeloma cell mass, stage 2 is intermediate tumor burden/cell mass, and stage 3 is a high tumor burden/cell mass.
  participants
    1 (a or b) | 0
    2a | 3
    2b | 1
    3a | 1
    3b | 0
International Staging System Classification [Number; unit: participants] — Stage I: β2M < 3.5 mg/l and serum albumin ≥3.5 g/100 ml (median survival 62 months); stage II, neither stage I nor stage III (median survival 44 months) and stage III β2M ≥5.5 mg/l (median survival 29 months)
  participants
    I | 0
    II | 3
    III | 2
Immunoglobulins [Number; unit: participants]
  IgG lambda Myeloma | 2
  Free Kappa light Chain Myeloma | 3

OUTCOME MEASURES:

1. Primary Outcome: Effect of Drug Combination on Multiple Myeloma
Description: The maximum response for all patients that were treated on study. Maximum response was assessed using the International myeloma working group (IMWG) guidelines for response. http://imwg.myeloma.org/international-myeloma-working-group-imwg-uniform-response-criteria-for-multiple-myeloma/
Time Frame: The best response for all patients at any point were assessed for patients that were treated on study, from start of treatment up to 20 weeks
Measure: Number; unit: participants
Arm/Group | DexTR (All Patients)
Number analyzed (Participants) | 5
participants
  partial response (PR) | 2
  minimal response (MR) | 1
  progression of disease | 2

ADVERSE EVENTS:
Arm/Group | DexTR (All Patients)
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DexTR (All Patients) (N=5)
sepsis (Infections and infestations) | 1
Fever (Infections and infestations) | 1
Cardiac Arrythmia (Cardiac disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to lack of sufficient accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less